CLINICAL TRIAL: NCT06094322
Title: Advanced DL-based T2w and DWI MR Sequences for Prostate Imaging
Brief Title: Evaluation of Rapid T2-weighted and DWI MR Sequences Reconstructed by Deep Learning for Prostate Imaging
Acronym: DLRPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2022_843_0108
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: T2 FSE; T2 DLR; diffusion DWI; diffusion DLR; Deep Learning Prostate cancer; PIRADS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MR prostate exam — Subjects will lie in supine position. The systematic use of a headset will reduce the acoustic noise inherent to the machine. We are going to carry out the standard MR prostate protocol which patients usually benefit from in clinical routine. This protocol consists of morphological sequences (T2 weighting with spin echo readout), Diffusion MR and dynamic contrast-enhanced sequences. We will then perform an additional faster enhanced T2-weighting SE and DWI sequences combined with Deep Learning reconstruction

SUMMARY:
MR prostate exam is essential for the diagnosis, workup and follow-up of prostate cancer. It allows to detect subclinical prostate cancer following an increase in the level of PSA. The investigators can score the lesion according to the PIRADS classification and obtain an estimate of lesion malignancy. To perform this classification, T2 and DWI sequences are essential.

Detection and characterization of malignant lesion is important to address appropriate patient care pathway. The purpose of this project is to evaluate novel deep learning (DL) T2-weighted TSE (T2DL) and Diffusion (DWIDL) sequences for prostate MR exam and investigate its impact on diagnostic, examination time, image quality, and PI-RADS classification compared to standard T2-weighted TSE (T2S) and standard Diffusion (DWIS) sequences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Healthy subject without history of hepatic disease
* Patient addressed for an prostate MRI
* Ability to give consent

Exclusion Criteria:

* claustrophobia,
* major obesity (>140 kg),
* Patient under guardianship or curators
* Age < 18 years,
* Women,
* History of prostatectomy or irradiation of the prostate
* any contraindication to MRI exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Change in number of suspicious nodule prostate detection before and after rapid T2-weighted | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No